CLINICAL TRIAL: NCT05300945
Title: HIPEC Combined Gastrectomy in Patients With Advanced Gastric Cancer Received Neoadjuvant Chemotherapy
Status: Not yet recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Zhixin Cao (Other)
Responsible Party: Sponsor-Investigator, Zhixin Cao, Prof, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TJ_HIPEC-01
Record Dates: First submitted 2022-03-20; First posted 2022-03-29 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: Gastric Cancer; Peritoneal Metastases
MeSH Terms: conditions — Stomach Neoplasms | interventions — Hyperthermic Intraperitoneal Chemotherapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (No Intervention)
- HIPEC (Experimental)
  Interventions: Combination Product: HIPEC

INTERVENTIONS:
Combination Product: HIPEC — HIPEC after gastrectomy with D2 local lymph node dissection.
  Arms: HIPEC

SUMMARY:
Patients with stage cT3-4N+M0 gastric cancer were recommended to receive neoadjuvant chemotherapy before radical surgery in terms of the eradication of micrometastasis in addition to local control, higher compliance with intensive chemotherapy, and avoidance of futile surgery by detection of initially invisible distant metastasis after rapid disease progression. However, in some studies, gastrectomy followed by neoadjuvant chemotherapy failed to demonstrate survival benefits for these patients. And peritoneal recurrence was the most common and devastating reason. Hyperthermic intraperitoneal chemotherapy (HIPEC) was introduced for peritoneal cancer last century. A few studies suggested HIPEC could improve prognosis in patients with limited peritoneal metastasis from various cancer. In summary, we conducted this study to confirm the efficacy and safety of HIPEC after gastrectomy in patients with advanced gastric cancer received neoadjuvant chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* histologically proven adenocarcinoma of stomach
* stage cT3-4N+M0
* no involvement of esophagus > 3 cm
* ECOG (Eastern Cooperative Oncology Group) : 0~1
* no previous chemotherapy or radiotherapy for any malignancy
* no previous surgery for GC excluding endoscopic mucosal resection or endoscopic submucosal dissection
* Signed the Informed Consent Form

Exclusion Criteria:

* Serious diseases that are difficult to control
* Severe hepatic and renal dysfunction
* Abnormal coagulation
* The presence of other serious physical or mental illness or laboratory abnormalities may increase the risk of participating in the study, or interfere with the results of the study, as well as the patients who the investigator believes are not suitable for participating in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Peritoneal recurrence | 3 years
OS | 3 years
  overall survival

SECONDARY OUTCOMES:
DFS | 3 years
  disease free survival
Adverse Events | 3 years
  Number and degree of Adverse Events

IPD SHARING:
Plan to Share IPD: Yes
All IPD that underlie results in a publication.
Supporting Information: Study Protocol, CSR
Time Frame: For 1 year after publishing the results in a journal.